CLINICAL TRIAL: NCT04992208
Title: Safety Observation of the Inactivated SARS-CoV-2 Vaccine (Vero Cell) in Population Aged 3~17 Years : A Multicenter,Open-label Study
Brief Title: Safety of an Inactivated SARS-CoV-2 Vaccine for Prevention of COVID-19 in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4008
Record Dates: First submitted 2021-08-02; First posted 2021-08-05 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): All of the participants(N=33000) will receive two doses inactivated SARS-CoV-2 vaccine . Vaccine will given by intramuscular injection on day 0 and day 28.
  Interventions: Biological: Experimental Group

INTERVENTIONS:
Biological: Experimental Group — SARS-CoV-2 Inactivated Vaccine 600SU inactivated virus in 0·5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac

SUMMARY:
This study is a multi-center and open design, phase Ⅳ clinical trial of an inactivated SARS-CoV-2 vaccine (CoronaVac) manufactured by Sinovac Research and Development Co., Ltd.The purpose of this study is to evaluate the safety of the SARS-CoV-2 Inactivated vaccine in population aged 3~17 years and in people with pre-existing disease to provide reference for improving the immunization strategy of COVID-19 vaccine.

DETAILED DESCRIPTION:
This study is a multi-center and open design, phase Ⅳ clinical trial in population aged 3~17 years . The experimental vaccine will be manufactured by Sinovac Research and Development Co.,Ltd.The study is planned to be carried out in 11 provinces from August 2021 to December 2022, including Liaoning, Heilongjiang, Anhui, Fujian, Jiangxi, Hubei, Guangxi, Chongqing, Guizhou, Yunnan and Gansu. Each province will serve as a research center, and each research center will select the corresponding research site.A total of 33000 subjects including patients with pre-existing will be enrolled with 3000 for each research center, including 600 subjects aged 3~5years，1200 subjects aged 6~11 years,1200 subjects aged 12~17 years.

And subjects will receive two doses of vaccine on day 0 and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Have not received any COVID-19 vaccine in the past or at least one dose of CoronaVac manufactured by Sinovac Research and Development Co.,Ltd;
* Population aged 3~17 years ;
* The subjects can understand and voluntarily sign the informed consent form and participate in the follow-up;

Exclusion Criteria:

* History of severe allergy to the vaccine such as acute allergic reaction,angioedema and dyspnea ;
* Severe neurological disease such as Myelitis transverse,Guillain-Barre Syndrome and demyelinating disorders;
* Acute disease,acute onset of chronic disease and severe chronic diseases.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31041 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Safety index 1-incidence of adverse reactions | Within 0~7 days after each dose
  Incidence rate of adverse reactions within 0~7 days after each dose in all populations.

SECONDARY OUTCOMES:
Safety index 2-incidence of adverse reactions | Within 0-28 days after each dose vaccination
  Incidence rate of adverse reactions within 0~28 days after each dose in all populations
Safety index 3-incidence of adverse reactions | Within 0~7 days after each dose vaccination
  Incidence of adverse reactions within 0~7 days after each dose in each age group
Safety index 4-incidence of adverse reactions | Within 0~28 days after each dose vaccination
  Incidence rate of adverse reactions within 0~28 days after each dose in each age group
Safety index 5-incidence of adverse reactions | Within 0~7 days after each dose vaccination
  Incidence of adverse reactions within 0~7 days after each dose in the population with pre-existing disease.
Safety index 6-incidence of adverse reactions | Within 0~28 days after each dose vaccination
  Incidence of adverse reactions within 0~28 days after each dose in the population with pre-existing disease.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Liu, Doctor, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention; Xing Fang, Principal Investigator — Liaoning Provincial Center for Disease Control and Prevention; Zhaodan Sun, Principal Investigator — HeilongjiangProvincial Center for Disease Control and Prevention; Fubing Wang, Principal Investigator — Hefei Provincial Center for Disease Control and Prevention; Dongjuan Zhang, Principal Investigator — Center for Disease Control and Prevention, Fujian; Shicheng Guo, Principal Investigator — Jiangxi Provincial Center for Disease Control and Prevention; Yeqing Tong, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention; Qiuyun Deng, Principal Investigator — Guangxi Center for Disease Control and Prevention; Qing Wang, Principal Investigator — Chongqing Center for Disease Control and Prevention; Ruizhi Zhang, Principal Investigator — Guizhou Provincial Center for Disease Control and Prevention; Xiaoshu Zhang, Principal Investigator — Gansu Provincial Center for Disease Control and Prevention
Locations (1):
- Yongping Center for Diseases Control and Prevention, Dali, Yunnan, China

REFERENCES:
- [Derived] Yang H, Li Z, Zhang R, Guo S, Wang B, Fang X, Zhang D, Zhang X, Tong Y, Wang Q, Deng Q, Sun Z, Liu X, Gao Y. Safety of primary immunization using inactivated SARS-CoV-2 vaccine (CoronaVac(R)) among population aged 3 years and older in a large-scale use: A multi-center open-label study in China. Vaccine. 2023 Feb 10;41(7):1354-1361. doi: 10.1016/j.vaccine.2023.01.020. Epub 2023 Jan 13. PMID 36658045